CLINICAL TRIAL: NCT03784326
Title: Phase I/II Study of Perioperative Chemotherapy Plus Immunotherapy Followed by Surgery in Localized Esophageal and Gastroesophageal Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0678; NCI-2018-02828 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0678 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-12-13; First posted 2018-12-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage II Esophageal Adenocarcinoma AJCC v8; Clinical Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IIA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IIB Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IC Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IC Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage II Esophageal Adenocarcinoma AJCC v8; Pathologic Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage III Esophageal Adenocarcinoma AJCC v8; Pathologic Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8
MeSH Terms: interventions — atezolizumab; Fluorouracil; dehydroftorafur; Oxaliplatin; Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1-Atezolizumab combination with Oxaliplatin and 5-fluorouracil (5-FU) (Experimental): The combination of Atezolizumab with Oxaliplatin and 5-Fluorouracil IV on Days 1 and 15 of each 28-day cycle for total of 6 doses followed by surgery followed by Atezolizumab on Day 1 of each 21-day cycle for total of 24 weeks
  Interventions: Drug: Atezolizumab; Procedure: Conventional Surgery; Drug: Fluorouracil; Drug: Oxaliplatin
- Cohort 2- Atezolizumab plus and Tiragolumab with Oxaliplatin and 5-fluorouracil (5-FU) (Experimental): The combination of Atezolizumab + Tiragolumab with Oxaliplatin and 5-Flourouracil IV on Days 1 and 15 of each 28-day cycle for total of 6 doses followed by surgery followed by Atezolizumab + Tiragolumab on Day 1 of each 21-day cycle for a total of 48 weeks.
  Interventions: Drug: Atezolizumab; Procedure: Conventional Surgery; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Tiragolumab

INTERVENTIONS:
Drug: Atezolizumab — Given IV (vein)
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Procedure: Conventional Surgery — Undergo surgical resection
Drug: Fluorouracil — Given IV (vein)
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Oxaliplatin — Given IV (vein)
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Drug: Tiragolumab — Given IV (vein)
  Arms: Cohort 2- Atezolizumab plus and Tiragolumab with Oxaliplatin and 5-fluorouracil (5-FU)

SUMMARY:
To learn if atezolizumab in combination with oxaliplatin and 5-fluorouracil (5-FU), when given before surgery, can help to control esophageal and/or gastroesophageal cancer. To learn if adding tiragolumab to the above drug combination can help to control the disease.

DETAILED DESCRIPTION:
Primary Objectives:

* Atezolizumab +/- tiragolumab in combination with oxaliplatin and 5-fluorouracil (modified FOLFOX) therapy in the neoadjuvant setting will achieve a pathological complete response of approximately 20% in patients with localized esophageal and gastroesophageal (GEJ) adenocarcinoma.

Secondary Objectives:

* To evaluate safety and toxicity profile of intravenous Atezolizumab +/- Tiragolumab in combination with Oxaliplatin and 5-FU chemotherapy as neoadjuvant treatment for resectable esophageal or GEJ adenocarcinoma.
* To assess the efficacy of the combination by tumor regression grade scoring in the surgical specimen.
* To assess the overall safety and tolerability of adjuvant Atezolizumab +/- Tiragolumab in subjects with resected esophageal and GEJ cancer
* To evaluate disease free survival (DFS) and overall survival (OS) in cohort 1 and cohort 2
* To explore changes in tumor stroma profile before and after immunotherapy in combination with chemotherapy

ELIGIBILITY:
Inclusion Criteria (cohort 1 and cohort 2)

* Signed Informed Consent Form
* Age ≥ 18 years at time of signing Informed Consent Form
* Ability to comply with the study protocol, in the investigator's judgment
* Histologically or cytologically confirmed esophageal or gastroesophageal type I or II adenocarcinoma
* No prior therapy including chemotherapy or radiation therapy.
* Patients with T1N1, and T2-3 with any N will be eligible.
* ECOG Performance Status of 0-1
* Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of study treatment:

  * ANC ≥ 1.5 x 109/L (1500/L) without granulocyte colony-stimulating factor support
  * Lymphocyte count ≥ 0.5 x 109/L (500/L)
  * Platelet count ≥ 100 x 109/L (100,000/L) without transfusion
  * Hemoglobin ≥ 90 g/L (9 g/dL) Patients may be transfused to meet this criterion.
  * AST, ALT, and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN)
  * Serum bilirubin ≤ 1.5 x ULN with the following exception:

Patients with known Gilbert disease: serum bilirubin level ≤ 3 x ULN

* Serum creatinine ≤ 1.5 x ULN [or] Creatinine clearance ≥ 70 mL/min (calculated using the Cockcroft-Gault formula)}
* Serum albumin ≥ 25 g/L (2.5 g/dL)
* For patients not receiving therapeutic anticoagulation: INR and aPTT ≤ 1.5 x ULN

  * For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
  * Medically fit for surgery based on surgeon's assessment.SAE
  * No supraclavicular, or para-aortic nodal enlargement unless biopsy negative.
  * Male or Female but both sexes must practice adequate contraception while on therapy. (please see required contraception below)
  * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) at screening, within 14 days prior to initiation of study treatment. Women must not be breastfeeding.
  * Availability of a representative tumor specimen that is suitable for determination of PDL-1 testing at MDA.

A formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or at least 10 slides containing unstained, freshly cut, serial sections should be submitted along with an associated pathology report prior to study enrollment. If <10 slides are available, the patient may still be eligible for the study, after principal investigator approval has been obtained. For Cohort 1: If archival tumor tissue is unavailable or is determined to be unsuitable for required testing, tumor tissue must be obtained from a biopsy performed at screening. Refer to Section 4.5.6 for additional information on tumor specimens collected at screening.

Options for female contraception

For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive, and agreement to refrain from donating eggs, as defined below:

Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the last dose of Atezolizumab, 90 days after the final dose of Tiragolumab, 4-9 months after the final dose of oxaliplatin and 6 months after the final dose of 5-FU. Women must refrain from donating eggs during this same period. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state ( 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

Hormonal contraceptive methods must be supplemented by a barrier method. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Options for contraception in male patients with pregnant female partners and/or with female partners of childbearing potential. "Recommendations related to contraception and pregnancy testing in clinical trials" and the Roche White Paper regarding contraception for males in clinical trials. Atezolizumab +/- Tiragolumab does require male contraception or condom use; guidelines below apply to other protocol-mandated study treatments.

• For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of 1% per year during the treatment period and for for 90 days after the final dose of tiragolumab, 6 months after the final dose of oxaliplatin and 5-FU to avoid exposing the embryo. Men must refrain from donating sperm during this same period.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria (cohort 1 and cohort 2)

* Patients with T1aN0, T4b, or metastatic cancer will be excluded.
* Squamous cell carcinoma histology
* Invasion into nearby organs (T4b) with or increased risk for fistula
* Significant comorbid conditions (defined as uncontrolled diabetes, active angina or heart failure, uncontrolled hypertension (>160 mmHg systolic or ≥100 mmHg diastolic) or increased risk of prolonged QTc (QTc > 500 ms), or active psychiatric condition that prevents consistent participation and compliance).
* More than grade 1 neuropathy.
* Unable to comprehend the requirements of the study or comply with it.
* Active bleeding from primary tumor requiring radiation therapy.
* History of leptomeningeal disease
* Uncontrolled tumor-related pain Patients requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.

Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.

* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Patients with indwelling catheters (e.g., PleurX) are allowed.
* Uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis with the following exceptions:

Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.

Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.

Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

* Rash must cover < 10% of body surface area
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids
* No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months

  * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
  * Positive HIV test at screening
  * Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test at screening Patients with a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test at screening, , an HBV DNA test should be performe before determining if patient is eligible for the study. (63)
  * Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test at screening The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
  * Active tuberculosis
  * Significant cardiovascular disease, such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
  * Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study
  * History of other malignancy within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS of > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
  * Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety.
  * Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
  * Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
  * Prior allogeneic stem cell or solid organ transplantation
  * Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment, within 90 days after the final dose of tiragolumab, or within 5 months after the final dose of atezolizumab
  * Positive Epstein-Barr virus (EBV) viral capsid antigen immunoglobulin M (IgM) test at screening An EBV PCR test should be performed as clinically indicated to screen for acute infection or suspected chronic active infection. Patients with a positive EBV PCR test are excluded.
  * Treatment with investigational therapy within 28 days prior to initiation of study treatment
  * Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, anti-TIGIT and anti-PD-L1 therapeutic antibodies
  * Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or five half-lives of the drug (whichever is longer) prior to initiation of study treatment
  * Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antiTNF- agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study, with the following exceptions:

Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator approval Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.

* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the oxaliplatin or 5-FU formulation
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months for atezolizumab+/- tiragolumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (PathCR) | Up to 3 years
  The optimum two-stage design proposed by Simon will be implemented. The PathCR rate will be estimated along with the exact 95% confidence interval.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | Up to 3 years
  The Kaplan-Meier method will be used to estimate the probabilities of DFS.
Overall survival (OS) | Up to 3 years
  The Kaplan-Meier method will be used to estimate the probabilities of OS.
Changes in tumor stroma profile after treatment | Baseline up to 3 years
  The changes in tumor stroma profile after treatment assessed through paired t-tests or Wilcoxon signed rank tests if normality assumption is not satisfied.
Incidence of toxicities defined as any treatment-related grade 3 or greater non-hematologic adverse events (AEs) determined by CTCAE version v 4.03. | From the start of study treatment up to 3 months
Tumor regression determined by CT or MRI | Baseline up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mariela Blum, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org